CLINICAL TRIAL: NCT02238288
Title: Randomized Clinical Trial to Verify the Effectiveness of Topical Aminocaproic Acid in the Prevention of Post-exodontic Bleeding in Patients on Anticoagulants
Brief Title: Randomized Clinical Trial With Aminocaproic Acid in the Prevention of Exodontic Bleeding in Anticoagulants Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Grupo de Estudos Multicentricos em Onco-Hematologia (Network)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AEAC2014
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Oral Hemorrhage
Keywords: anticoagulation; extraction; epsilon amino caproic
MeSH Terms: conditions — Oral Hemorrhage | interventions — Aminocaproic Acid; Lidocaine; Epinephrine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aminocaproic acid (Active Comparator): Crushed tablets inserted in the dental socket post-extraction
  Interventions: Drug: Aminocaproic acid; Drug: lidocaine and epinephrine; Drug: Paracetamol
- Routine care after dental extraction (Other): Chompret´s manoeuver, suture, surgical wound compression with gauze for 20 minutes
  Interventions: Other: Routine dental care; Drug: lidocaine and epinephrine; Drug: Paracetamol

INTERVENTIONS:
Drug: Aminocaproic acid — Crushed tablet in the dental socket
  Other Names: Ipsilon©
  Arms: aminocaproic acid
Other: Routine dental care — Chompret´s manoeuver, suture, surgical wound compression with gauze for 20 minutes
  Other Names: Routine procedures after dental extractions
  Arms: Routine care after dental extraction
Drug: lidocaine and epinephrine — 2%
Drug: Paracetamol — 750 mg

SUMMARY:
Patients using anticoagulants present an increased risk of bleeding when subjected to oral surgery. Suspending or reducing the oral anticoagulant dose to perform invasive procedures, may result in thromboembolic events, putting patients health in risk. Recent studies advocate the dental surgery treatment without suspending the anticoagulant therapy, since the values of the international normalized ratio (INR) are in acceptable therapeutic levels and local measurements are taken for the hemostasis control. The aim of this study is to compare the effectiveness use of intra-alveolar epsilon amino caproic acid (EACA) associated to daily rinses with the drug, with routine post-surgical procedures, to control the post-exodontic bleeding in anticoagulated patients. Patients will be referred by the anticoagulation clinic of the Clementino Fraga Filho University Hospital. Once the study criteria is met patients will be randomly allocated into two groups and subsequently subjected to clinical and periodontal examination, radiographic examination and pre-operative periodontal therapy. Laboratory tests (partial thromboplastic time, prothrombin time, international normalized ratio and platelet count) will be held on the day of the extraction. Patients in group 1 ( EACA ) will receive a paste composed of 01 macerated EACA tablet (500 mg), mixed with 0.9% saline solution in the alveolar socket, and routine post-operative care. Additionally, patients will perform oral rinses three times a day, on the first two post-operative days, with a solution from the macerated EACA 500mg tablet diluted in 2 spoons of filtered water. Patients allocated in group 2 (control) will receive routine post-operative care. Classification of immediate bleeding will be held by the professional, on the day of the surgery, immediately after the suture and twenty minutes later and the delayed bleeding, recorded by the patient through a daily questionnaire. The Statistical Package for the Social Sciences (SPSS)© (IBM, Chicago, USA) 20.0 is used as the database and the Chi-square, Kruskal-Wallis and Mann-Whitney tests will be applied to statistical analysis of the results.The study was approved by the ethical and research committee of the Clementino Fraga Filho University Hospital . All patients will sign a free consent and informed term.

DETAILED DESCRIPTION:
All patients will be submitted to clinical and radiographic examination. Once selected, patients will receive hygiene instruction and will be submitted to full mouth scaling one week before the procedure with an ultrasonic device (CavitronR - Dentsply). The random allocation of patients will obey the order obtained in the computerized program Allocation 1.0 Software© (Isfahan, Iran, 2004). All patients should have the prothrombin time (PT) and INR, active thromboplastin partial time (aTPT) and platelet counts tests on the day of surgery. Patients who present INR< 2.0 e > 4 will be assessed by the medical team about the possibility of change in the dose of medication to the surgical procedure. Patients with predisposing heart conditions the bacterial endocarditis will receive antibiotic prophylaxis as recommendations from American Association of Cardiology (AHA) of 2007. All extraction procedures will be performed by non-traumatic conventional surgical techniques, under local anesthesia (2% lidocaine and epinephrine 1: 100,000). Just one extraction will be performed in each surgical procedure, by the same surgeon. All patients will receive digital compression of socket with sterile gauze for 5 minutes (Chompret 's manoeuver) and suture with non-resorbable wire, silk 3.0 type . Everyone will receive the base analgesic prescription Paracetamol 750 mg (Tylenol© - Johnson & Johnson), 01 tablet every 6 hours, by oral administration, for control of postoperative pain. Patients are divided into two groups:

Group 1 (EACA) - patients will receive the intra-alveolar application of a 500 mg tablet of the epsilon-amino caproic acid (EACA - Ipsilon® - Nikko Brazil, RJ) crushed in 0.9% saline. Additionally, they will be instructed to rinse with 500mg EACA tablets macerated and diluted in 2 tablespoons of water three times a day, in the two days after the extraction.

Group 2 (control) - patients will receive routine postoperative care.

Classification of Bleeding will be performed by the professional on the day of surgery at two times: one time (immediately after extraction) and time 2 (after 20 minutes). The bleeding will be classified as follows:

* No bleeding
* Light bleeding - blood in saliva
* Moderate Bleeding - bleeding controlled with local measures
* Severe Bleeding - when surgical intervention is required

Late bleeding will be recorded by the patient through daily questionnaire. The bleeding will be classified as follows:

* No bleeding
* Blood stained saliva
* Bleeding that stopped after compression bandage and ice pack for 20 minutes
* Bleeding stopped only after professional intervention

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, use of warfarin sodium with or without anti-platelet aggregation, indicating simple extractions whose INR values are between 2.0 and 4.0 and that consent to participate in the study.

Exclusion Criteria:

* Patients with platelet count < 50,000 / mm3 Pregnant women or lactating Patients with hypersensitivity to the components of EACA. Patients with coagulopathies Patients who have impacted teeth, ankylosed or root morphological alterations that may complicate the procedure Patients who fail to submit laboratory and radiographic examinations necessary for the surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
bleeding post-exodontic | up to twenty minutes
  * No bleeding
  * Bleeding Light - blood in saliva
  * Moderate Bleeding - bleeding controlled with local measures
  * Severe Bleeding - when required surgical intervention and / or hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Clementino Fraga Filho University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil